CLINICAL TRIAL: NCT01843751
Title: Health Promotion and Public Safety: Community-based Collaborative Services to Addicted Offenders
Brief Title: Dane County Drug Court Study for Addicted Offenders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0226
Record Dates: First submitted 2013-04-17; First posted 2013-05-01 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2019-03

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician Office (Active Comparator): Buprenorphine/naloxone via physician office (B-PO) x 10 months
  Interventions: Drug: buprenorphine/naloxone
- Specialist Center (Experimental): Buprenorphine/naloxone via specialist center (B-SC) x 3 months followed by B-PO x 7 months. The specialist center in this trial will be a methadone clinic.
  Interventions: Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine/naloxone — Buprenorphine/naloxone (Suboxone) is considered a well-investigated, highly effective medication-assisted treatment for opiate dependence, but it may only be supervised through the few specialist treatment facilities in the state, or by physicians who have historically been less likely to offer this service. The effectiveness of community physician treatment supervision has not been tested for those in the criminal justice system.
  Other Names: Suboxone

SUMMARY:
The proposed work addresses critical health and public safety issues in the U.S. and in Wisconsin: the intersection of addiction and crime and the prevention of associated individual and public health complications. The results will provide justification for the expanded involvement of primary care in the treatment of substance-related disorders (opioid dependence in particular) and the prevention of their complications. As such, the project answers to federal calls for the expansion of substance abuse treatment into primary care settings and to objectives within the Alcohol and Drug Focus Area of Healthiest Wisconsin 2020.

DETAILED DESCRIPTION:
Addiction adversely affects individual and family well-being, public health, and public safety across the state of WI. Appropriate treatment can prevent myriad physical consequences of addiction, such as HIV, viral hepatitis, endocarditis, motor vehicle accidents and other trauma. Treatment to one addicted individual prevents 63 crimes per year-not including intimate partner and child abuse, which remain under-reported. An individual's contact with the WI criminal justice system constitutes a critical point for referral into supervised treatment to promote the recovery of the user and, hence, public health and safety. This project and related future work will help optimize prevention, intervention, and policy development targeting substance use, crime and related consequences. Specifically, the proposed work will 1) examine the impact of collaborative community treatment models involving generalist physician offices, specialist treatment facilities, and criminal justice, 2) examine HIV risk behaviors and their response to study conditions, and 3) disseminate results to state and national audiences to promote collaboration between criminal justice, specialist care, and generalist health care in reducing drug-related harms to individual and population health. There is a high prevalence of opiate dependence among the criminally involved. Buprenorphine/naloxone (Suboxone) is considered a well-investigated, highly effective medication-assisted treatment for opiate dependence, but it may only be supervised through the few specialist treatment facilities in the state, or by physicians who have historically been less likely to offer this service. The effectiveness of community physician treatment supervision has not been tested for those in the criminal justice system.

The proposed project seeks to test models to expand treatment access for substance dependent individuals. The project builds logically upon previous work by the PI. Substance dependent offenders are specifically chosen for investigation due to (1) the greater severity and prevalence of substance use problems and complications when compared to the more general adult substance-dependent population, (2) the impact of drug-related criminal behavior upon victims and upon the safety and well-being of our communities, and (3) the suitability of our team and community-based collaborators to conduct research with addicted offenders in order to promote individual recovery, public health, and public safety.

To contribute to knowledge regarding potential models for the expansion of treatment and supervision for substance dependent offenders, the current project and related future work will aim to:

1. Compare models of treatment involving (1) specialist-directed treatment followed by physician-office based treatment, and (2) physician-office-based treatment alone.
2. Determine if and to what degree a period of stabilization with specialist-directed treatment improves outcomes over physician-office-based treatment alone.
3. Clarify the optimal period of time for such a period of "specialist stabilization."

In this study, "stabilization" refers to a period of time at the front end of treatment during which the addicted offender participates in a more stringent set of supervisory conditions tied to their medication dispensing. This includes daily reporting for medication dosing and more frequent urine drug testing.

The primary study outcome will be time to commission of new crime. The primary outcome will be measured via the publicly available Wisconsin Circuit Court Consolidated Court Automation Program (CCAP) database. The Wisconsin Circuit Court Access website provides access to certain public records of the circuit courts of Wisconsin. The information displayed on the website is an exact copy of the case information entered into CCAP case management system by court staff in the counties where the case files are located. The court record summaries viewed are all public records under Wisconsin open records law and freely accessible to the public. The CCAP database will searched periodically for all enrolled study participants until data analysis has been complete.

Secondary outcomes include ongoing drug use as measured by urine drug testing, previously validated self-report measures; and treatment uptake and adherence. Secondary outcomes also include standardized measures of HIV risk behaviors, health services utilization, and cost benefit (societal perspective).

All subjects will be recruited via Journey Mental Health Center (formerly Mental Health Center of Dane County), which serves as the assessment unit for the Dane County Drug Treatment Court (DTC). This study will determine whether varying periods of initial stabilization in specialist treatment affects outcomes vs. physician-office treatment alone. The study will randomize 40 participants to one of 2 conditions characterized by the duration or lack of the "specialist stabilization period": 1) buprenorphine/naloxone via physician office (B-PO) x 10 months, or 2) buprenorphine/naloxone via specialist center (B-SC) x 3 months followed by B-PO x 7 months. Subjects will receive behavioral treatment and court supervision as usual. The primary outcome will be time to re-arrest/new crime. Secondary outcomes include ongoing drug use measured by 1) urine drug testing, and 2) validated self-report measures, treatment uptake and adherence, standardized measures of HIV risk behaviors, health services utilization, and cost benefit.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Drug Treatment Court
* diagnosis of opioid dependence using the Addiction Severity Index-Lite and diagnosis by clinical staff of referring units
* opioid positive urine drug screen at baseline
* women of childbearing potential who have a negative screening urine pregnancy test and are willing to use reliable birth control methods throughout the duration of the study.

Exclusion Criteria:

* pregnancy
* women who are currently breastfeeding
* complex psychiatric co-morbidity (e.g. suicidality, psychosis)
* complex medical co-morbidity (e.g. major cardiovascular, renal, or gastrointestinal/hepatic disease)
* or current pharmacotherapy with an agent which is contraindicated in combination with buprenorphine/naloxone according to drug labeling (
* Specific medical conditions, to be identified via initial medical history and examination, which would necessitate exclusion from study participation include: paralytic ileus, coronary artery disease or heart arrhythmia, recent head injury, obstructive sleep apnea, severe asthma or COPD, end-stage renal disease, or severe morbid obesity.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall T Brown, MD, PhD, Principal Investigator — University of Wisconsin, Department of Family Medicine
Locations (1):
- University of Wisconsin, Department of Family Medicine, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially 24 participants consented,but 3 did not receive intervention or provide data, so only 21 participants were analyzed out of 24 enrolled.
Period: Overall Study
Arm/Group | Physician Office | Specialist Center
Started | 11 | 10
Completed | 0 | 3
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician Office | Specialist Center | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 25 [17 to 43] | 22 [17 to 41] | 24 [17 to 43]
Sex: Female, Male [Count of Participants; unit: Participants] — One participant in "Specialist Center" arm did not provide Sex. Population: One participant in Specialist arm did not enter "Sex" information.
  Participants
    number analyzed (Participants) | 11 | 9 | 20
    Female | 4 | 3 | 7
    Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Crime
Description: The primary outcome will be measured via the publicly available Wisconsin Circuit Court Consolidated Court Automation Program (CCAP) database. The Wisconsin Circuit Court Access website provides access to certain public records of the circuit courts of Wisconsin. The information displayed on the website is an exact copy of the case information entered into CCAP case management system by court staff in the counties where the case files are located. The court record summaries viewed are all public records under Wisconsin open records law and freely accessible to the public. The CCAP database will searched periodically for all enrolled study participants until data analysis has been complete.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Office | Specialist Center
Number analyzed (Participants) | 11 | 10
Participants | 5 | 3

2. Secondary Outcome: Number of Days From Treatment Initiation to First Drug Use
Description: Number of days from treatment initiation to first drug use thereafter
Time Frame: 6 months
Measure: Mean (Full Range); unit: days
Arm/Group | Physician Office | Specialist Center
Number analyzed (Participants) | 11 | 10
days | 24 [0 to 182] | 15 [0 to 20]

3. Secondary Outcome: Initiation of Medication Assisted Treatment
Description: Initiation of medication assisted treatment (yes/no)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Office | Specialist Center
Number analyzed (Participants) | 11 | 10
Participants | 11 | 10

4. Secondary Outcome: Human Immunodeficiency Virus (HIV) Risk Behavior Assessment by Assessing Change in Risk Assessment Battery (RAB) Score
Description: The RAB is a self-administered, multiple choice questionnaire. It offers a quick and confidential assessment of both needle sharing practices and sexual activity associated with HIV transmission.
  The RAB is composed of 45 simple questions which uses discrete response. The questions have different numbers of items, and scores for a single question can range from 0 to 7, with higher values reflecting more instances of risk behavior. The RAB is scored by adding the values that correspond to the responses selected by the subject for the items. This total score is then divided by 40, the highest possible score for the overall instrument, yielding a score from 0 to 1.
  HIV risk behaviors will be assessed via score on the Risk Assessment Battery at baseline and month 6--difference between baseline and month 6.
Time Frame: baseline and 6 months
Population: Many subjects did not complete measurement at 6 months: 10 in physician office arm; 5 in specialist arm
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Physician Office | Specialist Center
Number analyzed (Participants) | 1 | 5
score on a scale | 0.01 [0.01 to 0.01] | 0.12 [0 to 0.19]

5. Secondary Outcome: Number of Emergency Room Visits
Description: Number of emergency room visits over 6 months
Time Frame: 6 months
Population: Many participants lost to follow up (9 in physician group, 5 in specialist group) who did not provide 6 month follow up data.
Measure: Mean (Full Range); unit: visits
Arm/Group | Physician Office | Specialist Center
Number analyzed (Participants) | 2 | 5
visits | 0 [0 to 0] | 0.2 [0 to 1]

ADVERSE EVENTS:
Arm/Group | Physician Office | Specialist Center
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes